CLINICAL TRIAL: NCT04883476
Title: A Prospective Study to Identify New "Omics" and Imaging Biomarkers of Chronic/Persistent Neck and Low Back Pain
Brief Title: Chronic Low Back Pain and Neck Pain Prospective Study
Status: Active, not recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Jason Pui Yin Cheung, Clinical Associate Professor, The University of Hong Kong
Other Study IDs: Study Protocol v. 1.0
Record Dates: First submitted 2021-04-26; First posted 2021-05-12 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Chronic Low Back Pain; Chronic Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tests for low density lipoprotein (LDL), high density lipoprotein (HDL), cholesterol counts, triglycerides, erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), metabolomics, glycomics, CCL5/CCL6 and adipokines.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic Low Back Pain and Neck Pain
  Interventions: Other: Observation study only

INTERVENTIONS:
Other: Observation study only

SUMMARY:
This prospective observation multifaceted study aims:

1. To perform a large prospective study and identify multiple "omics" biomarkers in chronic low back pain
2. To validate identified biomarkers for progression of acute to chronic low back pain
3. To validate identified biomarkers and test their heritability/validity in additional cohorts
4. To identify pathways and relevant individual variations for generation, propagation and subsidence of pain
5. To identify new imaging biomarkers related to chronic low back pain
6. To develop a registry of neck and low back pain subjects to help monitor the health-care management and utility to improve protocols and patient outcomes.

DETAILED DESCRIPTION:
This novel study aims to identify genetic variants associated with chronic low back pain as well as "omics and imaging biomarkers". To achieve this, we will link and relate clinical data (clinical and neurological signs leading to anatomical diagnosis plus a careful evaluation of inflammatory response of patient) to a multiple "omics" analysis in order to investigate promising biomarkers that could answer unmet needs: identification of predisposition to develop chronic low back pain, diagnosis and an objective measure of pain intensity in order to correlate to its pathophysiology, and validate predictors of response to specific (drug) treatments.

ELIGIBILITY:
Inclusion Criteria:

* Neck and/or low back pain
* New cases*
* Males and females
* 18 years or older
* Willing to participate in the study short- and long-term

Exclusion Criteria:

* Previous spine surgery
* Cognitively impaired
* Drug addiction
* Incarceration (prisoner)
* History of infections, tumors, chronic inflammation (e.g. rheumatoid arthritis, ankylosing spondylitis)
* Congenital/syndromal
* Pregnant females
* Diagnosed psychological impairment
* Inability to read or write

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were referred to the specialist orthopaedic clinic
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2015-05-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Radiographic assessment | Change up to 60-months follow-up
  assess the subjects' standing X-ray of the whole spine (AP and lateral) for the presence and extent of atherosclerosis, endplate thickening (sclerosis), vertebral osteophytes, limbus vertebrae, presence and categorization of vertebral subluxation (spondylolisthesis), additional spine-related deformities, spinal canal and vertebral body/foraminal dimensions, and static/dynamic spinal motion parameters and alignments. This will be done at interval follow-ups
MRI assessment | Change up to 60-months follow-up
  MRI:
  Sagittal T2W MRI whole spine and axial T1W MRI of lumbar spine will be assessed in all subjects. The radiographic events/outcomes of interest entailed the presence and extent of disc degeneration, disc bulges/herniations, Schmorl's nodes (endplate irregularities), high-intensity zones (HIZ), and bone marrow signal changes involving the endplate. Interval assessments will be made.

SECONDARY OUTCOMES:
Oswestry Disability index | Change to 60-months follow-up
  Questionnaire assessment: ODI is based on a 0-5 scale with 5 representing greatest disability. The index is calculated by dividing the summed score by the total possible score then multiplied by 100 as a percentage.
Neck disability index | Change to 60-months follow-up
  Questionnaire assessment: NDI assesses neck pain related disability. There are 10 items scored from 0-5 with maximum score of 50 indicating most severe pain.
Neck pain disability scale | Change to 60-months follow-up
  Questionnaire assessment: NPAD is a composite score of 20 items. Each score ranges from 0-5 with maximum score of 100 indicating maximal pain.
Depression-Anxiety Stress Scale | Change to 60-months follow-up
  Questionnaire assessment: DASS assesses symptoms based on a 4-point scale with subscales for depression, anxiety and stress. A range of 0-42 can be used with a higher score indicating worse severity.
SF-36 | Change to 60-months follow-up
  Questionnaire assessment: eight scaled score with weighted sums. Transformed to 0-100 scale, lower score means more disability.
VAS | Change to 60-months follow-up
  Questionnaire assessment for pain score. 0-10 with 10 being most severe.
Cholesterol assessment | Change to 60-months follow-up
  low density lipoprotein (LDL), high density lipoprotein (HDL), cholesterol counts, triglycerides
ESR | Change to 60-months follow-up
  Inflammatory marker via blood test
C-reactive protein | Change to 60-months follow-up
  Inflammatory marker via blood test

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Jason Cheung, Principal Investigator — The University of Hong Kong/ Queen Mary Hospital
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong